CLINICAL TRIAL: NCT01341366
Title: The Impact of Fast-track Perioperative Program on the Clinical and Immunological Outcomes After Laparoscopic Colorectal Surgery in Hong Kong Chinese Patients: A Prospective Randomized Trial
Brief Title: Fast-track Perioperative Program for Laparoscopic Colorectal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Simon S. M. Ng, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2008.552-T
Record Dates: First submitted 2011-04-20; First posted 2011-04-25 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Colorectal Cancer
Keywords: Laparoscopic surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fast-track perioperative program (Experimental)
  Interventions: Other: Fast-track perioperative program
- Traditional perioperative program (Active Comparator)
  Interventions: Other: Traditional perioperative program

INTERVENTIONS:
Other: Fast-track perioperative program — Preoperative counseling, no preoperative fasting, short-acting anesthetics, continuous infiltration of wound with local anesthetic agent, non-opioid pain management, the use of chewing gum, and early postoperative feeding and mobilization
  Arms: Fast-track perioperative program
Other: Traditional perioperative program — Preoperative fasting, standard anesthetic management with no intraoperative fluid restriction, opioid pain management, no chewing gum, feeding/mobilization according to attending surgeon
  Arms: Traditional perioperative program

SUMMARY:
Background:

Laparoscopic colorectal surgery has been shown by randomized trials to be associated with better short-term clinical outcomes when compared with open surgery. However, in a traditional perioperative care setting, the reduction in hospital stay following laparoscopic surgery in these trials was modest. Fast-track perioperative programs have been introduced in the West to optimize perioperative factors to reduce the physiological/psychological stress of open colorectal surgery. However, few studies have evaluated the impact of fast-track programs on the outcomes after laparoscopic colorectal surgery.

Objective:

To compare the clinical and immunological outcomes of Hong Kong Chinese patients undergoing laparoscopic surgery for colorectal cancer with a "traditional" vs. a "fast-track" perioperative program.

Design:

Prospective randomized trial.

Subjects:

One hundred and twenty-eight consecutive patients undergoing elective laparoscopic resection of non-metastatic colonic and upper rectal cancer will be recruited.

Interventions:

Patients will be randomized to a "traditional" or a "fast-track" perioperative program.

Outcome measures:

Primary outcome: total postoperative hospital stay, including hospital stay of patients who are readmitted within 30 days after surgery. Secondary outcomes: immunological parameters (including systemic cytokine response and cell-mediated immune function), morbidity and mortality, quality of life, and medical costs.

ELIGIBILITY:
Inclusion criteria:

* Consecutive patients undergoing elective laparoscopic resection of colonic and upper rectal cancer,
* Age of patients between 18 and 75 years
* Patients with American Society of Anesthesiologists grading I-II
* Patients with no severe physical disability
* Patients who require no assistance with the activities of daily living
* Informed consent available

Exclusion criteria:

* Patients undergoing laparoscopic low anterior resection with total mesorectal excision, abdominoperineal resection, or total/proctocolectomy
* Patients with planned stoma creation
* Patients undergoing emergency surgery
* Patients with known metastatic disease
* Patients with previous history of abdominal surgery
* Patients with known immunological dysfunction
* Patients who are taking steroids or immunosuppressive agents
* Patients with chronic pain syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2010-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Duration of hospital stay | Up to 1 month
  Total postoperative hospital stay, including hospital stay of patients who are readmitted within 30 days after surgery.

SECONDARY OUTCOMES:
Pain scores | Up to 1 week
  Pain scores on visual analogue scale (from 0 which implies no pain at all, to 100 which implies the worst pain imaginable)
Morbidity and mortality | Up to 1 month
Readmission rate | Up to 1 month
Quality of life | Up to 1 month
  Measured by SF-36, EORTC QLQ-C30 and QLQ-CR38 questionnaires
Direct/indirect medical costs and out-of-hospital economic costs | Up to 1 month
Systemic cytokine responses | Up to 1 week
  Blood levels of IL-1β, IL-6, and C-reactive protein
Lymphocyte subsets | Up to 1 week
  Using flow cytometer to determine lymphocyte subsets and NK cell counts (cells/uL)

CONTACTS AND LOCATIONS:
Overall Officials: Simon SM Ng, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, China

REFERENCES:
- See also: Related Info — http://www.surgery.cuhk.edu.hk